CLINICAL TRIAL: NCT06052111
Title: Dexmedetomidine Versus Fentanyl on Time to Extubation in Patients With Morbid Obesity Undergoing Laparoscopic Sleeve Gastrectomy: A Randamized Controlled Trial
Brief Title: Dexmedetomidine vs Fentanyl on Time to Extubation in Patients Undergoing Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Doha Mohammed Bakr, Assistant lecturer in Anesthesiology, Intensive care and Pain management, Faculty of Medicine, Helwan University, Qism Helwan Egypt., Helwan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 26-2020
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Dexmedetomidine; Fentanyl; Time to Extubation; Morbid Obesity; Laparoscopic Sleeve Gastrectomy
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group F (fentanyl group) (Experimental): Fentanyl (1 μg/kg) was given intravenously slowly over 60 seconds before induction of anesthesia as a loading dose followed by continuous infusion at a rate of (1μg/kg/hr) after intubation. It was stopped 10 minutes before the end of surgery.
  Interventions: Drug: Group F (fentanyl group)
- Group D (dexmedetomidine group) (Experimental): The patients were received a loading dose of dexmedetomidine (1 μg/kg) intravenously over 15 minutes before induction of anesthesia, followed by continuous infusion at a rate of (0.6 μg/ kg/ hr) after intubation and was stopped 10 minutes before the end of surgery.
  Interventions: Drug: Group D (dexmedetomidine group)

INTERVENTIONS:
Drug: Group F (fentanyl group) — Fentanyl (1 μg/kg) was given intravenously slowly over 60 seconds before induction of anesthesia as loading dose followed by continuous infusion at a rate of (1μg/kg/hr) after intubation and was stopped 10 minutes before the end of surgery.
  Arms: Group F (fentanyl group)
Drug: Group D (dexmedetomidine group) — The patients received loading dose of dexmedetomidine (1 μg/kg) (Precedex, Abbot Laboratories Inc., Abbot Park, IL, USA) intravenously over 15 minutes before induction of anesthesia followed by continuous infusion at a rate of (0.6 μg/ kg/ hr) after intubation and was stopped 10 minutes before the end of surgery.
  Arms: Group D (dexmedetomidine group)

SUMMARY:
This study aims to compare the efficacy of dexmedetomidine versus fentanyl during general anesthesia for patients with morbid obesity undergoing laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
The use of opioids in surgeries for patients with morbid obesity is controversial since they are known for having ventilatory depressing effects. Therefore, alternative analgesics are needed to improve anesthetic management for patients with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 50 years old.
* Both sexes.
* American Standards Association (ASA) physical status II - III.
* Body Mass Index (BMI) ≥ 35 kg/m2.

Exclusion Criteria:

* Allergy to α2 -adrenergic agonist.
* History of cardiac disease (uncontrolled hypertensive patient with blood pressure above 140/90, implanted pacemaker, poor cardiac function (ejection fraction< 50%), history of myocardial infarction, cerebral stroke, transient ischemic attack, or coronary artery disease with or without stents.
* Neuromuscular disease, liver disease (coagulopathy INR>1.5 or platelet count <100.000/μl), renal impairment (serum creatinine >1.2mg/dl, serum K >5.5mmol/l).
* Opioid medication within 24 hours before the operation.
* Respiratory diseases as COPD, uncontrolled asthmatic patients.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
The time for extubation | 30 minutes till end of surgery.
  Time from end of anesthesia till safe extubation of the patients

SECONDARY OUTCOMES:
Mean arterial blood pressure (MAP) | Intraoperatively.
  Mean arterial blood pressure will be recorded (baseline, after induction, after tracheal intubation, at trochers insertion, during insufflation, at regular intervals throughout the surgery (every 5 minutes) until the end of surgery.
Heart rate (HR) | Intraoperatively
  Heart rate will be recorded (baseline, after induction, after tracheal intubation, at trochers insertion, during insufflation, at regular intervals throughout the surgery (every 5 minutes) until the end of surgery.
Incidence of hypotension | Intraoperatively
  Mean arterial blood pressure (MAP)<60mmHg. Ephedrine (5 mg) and 250 ml fluid bolus will be given if MAP < 60 mmHg or decrease 20% of the baseline value.

CONTACTS AND LOCATIONS:
Locations (1):
- Helwan University, Helwan, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year
Access Criteria: The data will be available upon a reasonable request from the corresponding author.